CLINICAL TRIAL: NCT02915081
Title: Blue Light Therapy for Liver Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low anticipated recruitment
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Allan Tsung, Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO13080427
Record Dates: First submitted 2016-09-10; First posted 2016-09-26 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Acute Kidney Injury; Liver Injury; Inflammation
MeSH Terms: conditions — Acute Kidney Injury; Inflammation | interventions — Blue Light

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue light (Experimental): Subjects will be exposed to 24 hours of bright (1700 lux) blue (peak 442 nm) spectrum light the day prior to operative intervention and for the 24 hours after the operative intervention.
  Interventions: Other: Blue light
- Ambient light (No Intervention): Subjects will be exposed preoperatively to the lighting conditions of their living environment and postoperatively to the standard, white fluorescent lighting environment of the hospital.

INTERVENTIONS:
Other: Blue light — Illumination: High illumination lighting will be instituted with a Day*Light Classic Light (Uplift Technologies, Dartmouth, NS)
  Blue wavelength: Each subject will be fitted with blue filtered goggles (Lee Filters, Burbank, CA). These goggles ensure the transmission of a bright (1700 lux) blue (peak 442 nm) spectrum light when the subject is within 12 inches.
  Photoperiod: A 24-hour photoperiod will be used that commences at 0800 the morning prior to surgery and continues for 24 hours. To account for potential variability in the exposure of interest, each subject will complete a diary to catalogue duration and distance of light exposure. Postoperatively the same photoperiod will be instituted and continued for one 24 hour period.
  Arms: Blue light

SUMMARY:
The investigators hypothesize that subjects undergoing liver resection and who are exposed preoperatively to high illuminance blue spectrum light will exhibit reduced organ injury, specifically liver dysfunction, than subjects exposed to standard ambient white fluorescent light.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 17 years
* undergoing right or left hepatic lobectomy

Exclusion Criteria:

* presence of acute traumatic brain injury
* blindness
* immunosuppression or immunocompromised condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline creatinine concentration at 24 hours after surgery | preoperatively and 24 hours after surgery
  a serum marker of acute kidney injury
Change from baseline alanine aminotransferase (ALT) concentration at 24 hours after surgery | preoperatively and 24 hours after surgery
  a serum marker of acute liver injury

SECONDARY OUTCOMES:
Change in serum cytokine concentrations at 24 hours after surgery | 24 hours after surgery
  serum will be analyzed for cytokines and inflammatory mediators
Ventilator-free days | for the duration of postoperative inpatient hospital stay up to 28 days
ICU length of stay | for the duration of postoperative inpatient hospital stay up to 28 days
renal replacement therapy | for the duration of postoperative inpatient hospital stay up to 28 days
Change in serum cytokine concentrations at 1 hour after surgery | 1 hours after surgery
  serum will be analyzed for cytokines and inflammatory mediators

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
This trial is a small pilot trial.